CLINICAL TRIAL: NCT01401062
Title: Fresolimumab and Radiotherapy in Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S11-00533; BC100481 (Other Grant/Funding Number: DOD)
Record Dates: First submitted 2011-07-20; First posted 2011-07-25 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic breast cancer; TGF-beta; fresolimumab; monoclonal antibody; radiation therapy; abscopal response
MeSH Terms: conditions — Breast Neoplasms; Camurati-Engelmann Syndrome | interventions — fresolimumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Fresolimumab 1 mg/kg) (Experimental): Fresolimumab is administered intravenously (i.v.) at a dose of 1 mg/kg on day 1 of weeks 0, 3, 6, 9 & 12 and radiation administered at 7.5 Gy/fraction in 3 fractions during weeks 1 (to lesion 1) and 7 (to lesion 2).
  Interventions: Drug: Fresolimumab; Radiation: Radiation Therapy
- Arm 2 (Fresolimumab 10 mg/kg) (Experimental): Fresolimumab is administered intravenously (i.v.) at a dose of 10 mg/kg on day 1 of weeks 0, 3, 6, 9 & 12 and radiation administered at 7.5 Gy/fraction in 3 fractions during weeks 1 (to lesion 1) and 7 (to lesion 2).
  Interventions: Drug: Fresolimumab; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Fresolimumab
  Other Names: GC1008
Radiation: Radiation Therapy

SUMMARY:
The purpose of this study is to test safety of combining fresolimumab and local radiotherapy and to see if the combination can achieve tumor regression.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven breast cancer, metastatic (persistent or recurrent).
* Failed ≥1 line of therapy (endocrine or chemotherapy) for metastatic disease.
* Min. 3 distinct metastatic sites, at least one measurable lesion which is at least 1 cm or larger in largest diameter.
* Must be ≥4 weeks since all of the following treatments (recovered from toxicity of prior treatment to ≤Grade 1, excluding alopecia):

  * major surgery;
  * radiotherapy;
  * chemotherapy (≥6 weeks since therapy if a nitrosourea, mitomycin, or monoclonal antibodies such as bevacizumab);
  * immunotherapy;
  * biotherapy/targeted therapies.
* >18 years of age.
* Life expectancy >6 months.
* Eastern Cooperative Oncology Group (ECOG) status 0 or 1.
* Adequate organ function including:

  * Hemoglobin ≥10.0g/dL, absolute neutrophil count (ANC) ≥1,500/mm3, and platelets ≥100,000/mm3.
  * Hepatic: Serum total bilirubin ≤1.5x upper limit of normal (ULN) (Patients with Gilbert's Disease may be included if total bilirubin is ≤3.0mg/dL), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤2.5xULN. If patient has known liver metastases, ALT and/or AST ≤5xULN are allowed.
  * Renal: creatinine clearance ≥60mL/min.
  * Prothrombin (PT) and partial thromboplastin times (PTT) <ULN.
* Negative for hepatitis viruses B and C unless consistent with prior vaccination or prior infection with full recovery.
* Patients of childbearing potential must agree to use effective contraception while on study, and for ≥3 months after last treatment.
* Understand and sign written informed consent document. No consent by durable power of attorney.

Exclusion Criteria:

* Second malignancy - unless following curative intent therapy, has been disease free for ≥2 years with probability of recurrence <5%. Curatively treated early-stage squamous cell carcinoma of the skin, basal cell carcinoma of the skin, or cervical intraepithelial neoplasia (CIN) are allowed.
* Concurrent cancer therapy.
* Uncontrolled central nervous system (CNS) metastases, meningeal carcinomatosis, malignant seizures, or disease that causes or threatens neurologic compromise (e.g. unstable vertebral metastases).
* History of ascites or pleural effusions, unless successfully treated.
* Organ transplant, including allogeneic bone marrow transplant.
* Immunosuppressive therapy including:

  * Systemic corticosteroid therapy, including replacement therapy for hypoadrenalism. Inhaled or topical corticosteroids are allowed (if therapy is <5 days and is limited to systemic steroids as antiemetics);
  * Cyclosporine A, tacrolimus, or sirolimus.
* Investigational agents within 4 weeks prior to study enrollment (≥6 weeks if treatment was long-acting agent such as monoclonal antibody).
* Significant or uncontrolled medical illness, e.g. congestive heart failure (CHF), myocardial infarction, symptomatic coronary artery disease, significant ventricular arrhythmias within the last 6 months, or significant pulmonary dysfunction. Patients with remote history of asthma or active mild asthma may participate.
* Active infection, including unexplained fever (>38.5°C).
* Systemic autoimmune disease (e.g. systemic lupus erythematosus, active rheumatoid arthritis).
* Known allergy to any component of GC1008.
* Active thrombophlebitis, thromboembolism, hypercoagulability states, bleeding, or anti-coagulation therapy (including anti platelet agents i.e. aspirin, clopidogrel, ticlopidine, dipyridamole, other agents inducing long-acting platelet dysfunction). Patients with history of deep venous thrombosis are allowed if treated, completely resolved, and no treatment for >4months.
* Calcium >11.0mg/dL (2.75mmol/L) unresponsive or uncontrolled in response to standard therapy (e.g. bisphosphonates).
* Patients who, in the opinion of the Investigator, have significant medical or psychosocial problems, including, but not limited to:

  * Other serious non-malignancy-associated conditions that may be expected to limit life expectancy or significantly increase the risk of SAEs;
  * Conditions, psychiatric, substance abuse, or other, that, in the opinion of the Investigator, would preclude informed consent, consistent follow-up, or compliance with any aspect of the study;
* Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Formenti, M.D., Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - New York University Langone Medical Center Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolchok JD, Hoos A, O'Day S, Weber JS, Hamid O, Lebbe C, Maio M, Binder M, Bohnsack O, Nichol G, Humphrey R, Hodi FS. Guidelines for the evaluation of immune therapy activity in solid tumors: immune-related response criteria. Clin Cancer Res. 2009 Dec 1;15(23):7412-20. doi: 10.1158/1078-0432.CCR-09-1624. Epub 2009 Nov 24. PMID 19934295
- [Derived] Formenti SC, Hawtin RE, Dixit N, Evensen E, Lee P, Goldberg JD, Li X, Vanpouille-Box C, Schaue D, McBride WH, Demaria S. Baseline T cell dysfunction by single cell network profiling in metastatic breast cancer patients. J Immunother Cancer. 2019 Jul 11;7(1):177. doi: 10.1186/s40425-019-0633-x. PMID 31296256
- [Derived] Sato M, Kadota M, Tang B, Yang HH, Yang YA, Shan M, Weng J, Welsh MA, Flanders KC, Nagano Y, Michalowski AM, Clifford RJ, Lee MP, Wakefield LM. An integrated genomic approach identifies persistent tumor suppressive effects of transforming growth factor-beta in human breast cancer. Breast Cancer Res. 2014 Jun 2;16(3):R57. doi: 10.1186/bcr3668. PMID 24890385

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 (Fresolimumab 1 mg/kg): Fresolimumab is administered intravenously (i.v.) at a dose of 1 mg/kg on day 1 of weeks 0, 3, 6, 9 & 12 and radiation administered at 7.5 Gy/fraction in 3 fractions during weeks 1 (to lesion 1) and 7 (to lesion 2).
  Fresolimumab
  Radiation Therapy
- Arm 2 (Fresolimumab 10 mg/kg): Fresolimumab is administered intravenously (i.v.) at a dose of 10 mg/kg on day 1 of weeks 0, 3, 6, 9 & 12 and radiation administered at 7.5 Gy/fraction in 3 fractions during weeks 1 (to lesion 1) and 7 (to lesion 2).
  Fresolimumab
  Radiation Therapy
Period: Overall Study
Arm/Group | Arm 1 (Fresolimumab 1 mg/kg) | Arm 2 (Fresolimumab 10 mg/kg)
Started | 11 | 12
Completed | 0 | 4 (At time of data entry, these 4 patients are still undergoing follow-up)
Not Completed | 11 | 8
Not completed — Death | 9 | 7
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (Fresolimumab 1 mg/kg) | Arm 2 (Fresolimumab 10 mg/kg) | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 7 | 16
  >=65 years | 2 | 5 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian or Pacific Islander | 1 | 3 | 4
  Black, not of Hispanic-American Origin | 3 | 0 | 3
  White, not of Hispanic-American origin | 6 | 8 | 14
  Other/Unknown | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Abscopal Response Rate
Description: Defined as the percentage of patients who have responses (complete or partial) outside the irradiated lesions. The abscopal response is assessed at 15 weeks, and confirmed minimum 4 weeks later. The abscopal response is evaluated based on immune-related response criteria (irRC) (Wolchok et al, 2009).
Time Frame: up to 20 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Fresolimumab 1 mg/kg) | Arm 2 (Fresolimumab 10 mg/kg)
Number analyzed (Participants) | 11 | 12
Participants | 11 | 12

ADVERSE EVENTS:
Arm/Group | Arm 1 (Fresolimumab 1 mg/kg) | Arm 2 (Fresolimumab 10 mg/kg)
Serious Adverse Events (participants affected / at risk) | 3/11 | 3/12
Other Adverse Events (participants affected / at risk) | 9/11 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (Fresolimumab 1 mg/kg) (N=11) | Arm 2 (Fresolimumab 10 mg/kg) (N=12)
atrial fibrillation (Cardiac disorders) | 2 | 0
Hypercalcemia (Endocrine disorders) | 1 | 1
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Dyspnea (Immune system disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cord compression (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (Fresolimumab 1 mg/kg) (N=11) | Arm 2 (Fresolimumab 10 mg/kg) (N=12)
hypercalcemia (Metabolism and nutrition disorders) | 1 | 1
Aspartate Aminotransferase Increased (Investigations) | 3 | 0
Alkaline Phosphate Increased (Investigations) | 2 | 0
Bilaterial Effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Cord compression (Nervous system disorders) | 1 | 0
Neuropathy (Nervous system disorders) | 1 | 0
Spinal Edema (Skin and subcutaneous tissue disorders) | 1 | 0
alanine aminotransferase (Investigations) | 1 | 0
Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Fatigue (General disorders) | 3 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
INR (Investigations) | 1 | 0
Neuropathy- Lower Extremities (Nervous system disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 1
Lower Sacral Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Abdominal Pain- Severe (Gastrointestinal disorders) | 1 | 0
Pain (under R breast) (Reproductive system and breast disorders) | 1 | 0
Elevated Bilirubin (Investigations) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Elevated Amylase (Investigations) | 1 | 0
Elevated Lipase (Investigations) | 1 | 0
Hepatic Encephalopathy (Nervous system disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oliguria (Investigations) | 1 | 0
Cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0
PTT (Investigations) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Elevated AST (Investigations) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No